CLINICAL TRIAL: NCT07260292
Title: Kefir Peptides Supplement for Inflammation, Oxidative Stress and Lipid Abnormalities in Chronic Kidney Disease Patients
Brief Title: KPs Supplement for Inflammation, Oxidative Stress and Lipid Abnormalities in CKD Patients.
Acronym: KPs; CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Chung Hsing University (Other)
Collaborators: Jen Ai Hospital (Unknown)
Responsible Party: Principal Investigator, Chuan -Mu Chen, Chair Professor, National Chung Hsing University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHP2201H04; 111-89 (Other Grant/Funding Number: Jen-Ai Hospital)
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease Stage 3; Chronic Kidney Disease Stage 4; Proteinuria
Keywords: Chronic kidney disease; Gut dysbiosis; Proteinuria; Kefir peptides,; Postbiotics
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, parallel study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and investigators were unaware of group assignment; placebo was identical in appearance to study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KEFPEP® (Experimental): Powder (directly take the powder with appropriate amount of warm water)
  Interventions: Dietary Supplement: KEFPEP®
- Placebo (Placebo Comparator): Powder (directly take the powder with appropriate amount of warm water)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: KEFPEP® — oral administration at a daily dosage of 2.4 grams for 12 weeks
  Arms: KEFPEP®
Dietary Supplement: Placebo — using regular yogurt powder as a substitute for KPs
  Arms: Placebo

SUMMARY:
This clinical investigation is designed to evaluate the potential therapeutic effects of kefir peptides as an adjunct intervention for chronic kidney disease (CKD) and clinical proteinuria. Patients diagnosed with stage 3 or 4 CKD will receive a three-month course of kefir peptide supplementation. Throughout the intervention period, the investigator will monitor renal function markers (blood urea nitrogen, serum creatinine), proteinuria (urine protein-to-creatinine ratio), inflammatory indicators (high-sensitivity C-reactive protein), and additional biochemical parameters relevant to CKD progression.

DETAILED DESCRIPTION:
Background and Aim Chronic kidney disease (CKD) represents a substantial global public health burden, with prevalence rising due to population aging and an increased incidence of systemic conditions such as hypertension, diabetes mellitus, metabolic syndrome, and chronic exposure to nephrotoxic agents. Accumulation of uremic toxins in CKD contributes to gut dysbiosis, systemic inflammation, accelerated renal functional decline, and heightened cardiovascular risk.

Probiotics and postbiotics have been evaluated as potential adjunct therapies to slow CKD progression; however, conclusive evidence supporting their clinical effectiveness remains limited. Kefir peptides (KPs) contain bioactive constituents with documented antioxidant, antidiabetic, antithrombotic, antibacterial, anti-osteoporotic, and immunomodulatory properties. Based on these characteristics, KPs may offer therapeutic benefits in modulating renal function, systemic inflammation, and uremic toxin burden in individuals with advanced CKD.

The current investigation aims to examine the effects of kefir peptides on renal function and clinical proteinuria, and to explore possible mechanistic pathways contributing to these outcomes.

Methods A total of 165 participants were enrolled: 83 in the placebo group and 82 in the kefir peptide group. All participants consumed the assigned kefir formulation twice daily for three months. Blood and urine biochemical assessments were conducted at baseline (week 0), week 4, and week 12. Serum high-sensitivity C-reactive protein (hs-CRP), indoxyl sulfate (IS), and p-cresyl sulfate (PCS) levels were measured at baseline and at week 12. All study procedures and monitoring activities were performed by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age: 30-82 years of age
* Chronic kidney disease stage 3 and 4
* Sign informed consent

Exclusion Criteria:

* Acute illness
* Pregnancy
* Aboriginal descent

Ages: 30 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in renal function biomarker( BUN & Cr) | Baseline to 12 weeks
Change in urine protein-to-creatinine ratio (UPCR) | Baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: YU-HSIEN LIU, Master, Study Director — Jen Ai Hospital
Locations (1):
- Jen-Ai Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns regarding patient privacy and confidentiality. Only de-identified and aggregated data will be included in future publications or presentations.

REFERENCES:
- [Background] Liu YH, Chen YH, Ko CH, Kuo CW, Yen CC, Chen W, Chong KY, Chen CM. SOD3 and IL-18 Predict the First Kidney Disease-Related Hospitalization or Death during the One-Year Follow-Up Period in Patients with End-Stage Renal Disease. Antioxidants (Basel). 2022 Jun 18;11(6):1198. doi: 10.3390/antiox11061198. PMID 35740095